CLINICAL TRIAL: NCT07270900
Title: A Mindfulness-based Intervention for Adolescents With Prediabetes or Type 2 Diabetes
Acronym: L2BT2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tamara S. Hannon, Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21496
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes; Prediabetes
Keywords: mindfulness based intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Learn to Breathe Group Program (Experimental): All study participants take part in the L2B MBI
  Interventions: Procedure: Mindfulness Based Group

INTERVENTIONS:
Procedure: Mindfulness Based Group — L2B is a manualized 12-week curriculum that teaches a variety of mindfulness skills including breath awareness, body scanning, mindful eating, sitting meditation, loving kindness practice, and mindful movement. Weekly group sessions will last 45-60 minutes. Participants will be invited to engage in daily practice of mindfulness skills (home practice).

SUMMARY:
The purpose of this study is to conduct a mindfulness-based intervention for adolescents referred for prediabetes or type 2 diabetes treatment to 1) evaluate feasibility and acceptability of the intervention for future research and clinical use and 2) explore secondary health outcomes related to diabetes prevention and care.

DETAILED DESCRIPTION:
Background and Rationale Mindfulness-based interventions (MBI) may offer additional benefits to traditional health care for youth living with prediabetes or T2D. MBIs teach skills to increase present moment attention and adopt a nonjudgmental attitude towards one's experience which can foster healthy stress coping behaviors and greater self-regulation; both of which are associated with improved diabetes self-care behaviors. MBIs were introduced to the clinical population in the 1970's and have been translated for a variety of populations and health conditions including diabetes. MBIs may be a promising complementary approach for T2D prevention and treatment in youth, and thus, warrant further investigation.

Specific Aims Aim 1: Pilot test the feasibility and acceptability of a mindfulness-based intervention in adolescents with prediabetes or type 2 diabetes.

Aim 2: Explore secondary physical and mental health outcomes of the study cohorts.

Enrollment The investigators aim to recruit 50 individuals with the goal of at least 20 participants to complete the study (two groups of 10 participants).

Recruitment Sites: Diabetes care providers see patients in an outpatient setting at Riley Specialty Care at IU Health Methodist in Indianapolis, Indiana. Additional outreach clinics available for participant recruitment include Riley Specialty Care at Riley Outpatient Center, IU North, Bloomington, Fort Wayne, and South Bend.

Study Procedures Following enrollment, participants will complete baseline surveys and begin attending the 12-week MBI. Participants will complete surveys following completion of the MBI and at the 12-month follow up.

Intervention The MBI will be conducted in a virtual group setting by Zoom, with a target size of 8-12 participants. Groups may vary in size based on session attendance. The MBI will follow the Learning to BREATHE (L2B) curriculum. L2B is a manualized 12-week curriculum that teaches a variety of mindfulness skills including breath awareness, body scanning, mindful eating, sitting meditation, loving kindness practice, and mindful movement. Weekly group sessions will last 45-60 minutes. Participants will be invited to engage in daily practice of mindfulness skills (home practice). This study includes a post-intervention group guided interview at 12-weeks. The facilitator will ask the group for feedback about the intervention with the following questions: 1) What did you like about participating in this study? 2) What did you dislike about participating in this study? 3) What were your expectations from participating in this study? 4) Were those expectations met?

The investigators will describe the results of participants using quantitative data (results of surveys and numerical clinical information from HbA1c and BMI) and qualitative data (results from interviews).

This study will be important to serve as the foundation for a fully powered clinical trial of MBI in type 2 diabetes and prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years
* Referred to clinic for treatment of prediabetes or type 2 diabetes
* English speaking

Exclusion Criteria:

* • Diagnosed cognitive disabilities

  * Inability to attend visits due to individual schedules

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Participation | 3 months
  Study Participation Rate: Number of participants who consented to take part in the study divided by the number of patients approached. We will also document reasons for refusal to participate in the study.
Acceptability | 12 months
  L2B Program Questionnaires
  Post-study guided interview:
  1. What did you like about participating in this study?
  2. What did you dislike about participating in this study?
  3. What were your expectations from participating in this study?
  4. Were those expectations met?
Recruitment | 3 months
  Time to Recruit: Time required to attain the needed sample for each recruitment wave
Attendance | 4 months
  Attendance: Attendance at each intervention session will be recorded.
Retention | 12 months
  Study Retention Rate: Number of participants in a study arm who remain in the study and maintain communication with study staff (regardless of session attendance) divided by the number of participants enrolled in the study.
Completion | 12 months
  Study Completion Rate: Number of participants who complete all assessments divided by the number of participants enrolled in the study arm.
Data Completeness | 12 months
  Data Completeness: Percentage of questionnaires/study measures completed.

SECONDARY OUTCOMES:
Height from electronic medical record | 12 months
  Height in centimeters from electronic medical record
HbA1c from electronic medical record | 12 months
  HbA1c from electronic medical record
Weight from the electronic medical record | 12 months
  Weight in kilograms from the electronic medical record

OTHER OUTCOMES:
Anxiety symptoms | 12 months
  Screen for Childhood Anxiety Related Emotional Disorders (SCARED-5); 5 items; A score of ≥3 indicates the possibility of anxiety.
Depression symptoms | 12 months
  Depression-Pediatric Item Bank (PROMIS) - 14 items; A T-score of 50 is the mean; higher scores indicate more depressive symptoms.
Perceived Stress Scale | 12 months
  Perceived Stress Scale (PSS-10): 10 items; score 0-40; higher scores indicate more stress.
Health-related quality of life | 12 months
  Peds QL Generic Core Scales: 23 Items; generic Core Scales scores are transformed on a scale from 0-100 with higher scores indicating higher health-related quality of life.
Mindful attention awareness | 12 months
  Mindful Attention Awareness Scale (MAAS); 15 items; higher scores indicate more mindful attention awareness.
Emotion regulation | 12 months
  Difficulties in Emotion Regulation Scale (DERS); 36 items; higher scores indicate more difficulties with emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara S Hannon, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Diabetes CLinic, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as the data for this study is strictly confidential.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT07270900/Prot_SAP_000.pdf